## **Informed Consent Form**

Winship3185-16: A Phase II Trial of Pembrolizumab (MK-3475) in Metastatic Cutaneous Squamous Cell Carcinoma

NCT Number: NCT02964559

Document IRB Approval Date: 9/11/2019



## You Are Being Asked to Be in a Research Study

## What Is a Research Study?

The main purpose of research studies is to gain knowledge. This knowledge may be used to help others. Research studies are not intended to benefit you directly, though some might.

## Do I Have to Do This?

No. Being in this study is entirely your choice. If you decide to join this study, you can change your mind later on and withdraw from the research study.

Taking part in a study is separate from medical care. The decision to join or not join the research study will not affect your status as a patient.

### What Is This Document?

This form is an informed consent document. It will describe the study risks, procedures, and any costs to you.

This form is also a HIPAA Authorization document. It will describe how your health information will be used and by whom.

Signing this form indicates you are willing to take part in the study and allow your health information to be used.

## What Should I Do Next?

- 1. Read this form, or have it read to you.
- 2. Make sure the study doctor or study staff explains the study to you.
- 3. Ask questions (e.g., time commitment, unfamiliar words, specific procedures, etc.)
- 4. If there will be medical treatment, know which parts are research and which are standard care.
- 5. Take time to consider this, and talk about it with your family and friends.

Version Date: 04/15/2019 IRB Form 01292016

Document Approved On: 9/11/2019

# Emory University Consent to be a Research Subject / HIPAA Authorization

<u>Title</u>: Winship 3185-16 A Phase II trial of pembrolizumab (MK-3475) in metastatic cutaneous (skin) squamous cell carcinoma

Principal Investigator: Ragini R. Kudchadkar, MD

Investigator-Sponsor: Ragini R. Kudchadkar, MD

**Study-Supporter:** Merck

#### Introduction

You are being asked to be in a medical research study. This form is designed to tell you everything you need to think about before you decide if you want to be a part of the study. It is entirely your choice. If you decide to take part, you can change your mind later on and withdraw from the research study. The decision to join or not join the research study will not cause you to lose any medical benefits. If you decide not to take part in this study, your doctor will continue to treat you.

## Before making your decision:

- Please carefully read this form or have it read to you
- Please listen to the study doctor or study staff explain the study to you
- Please ask questions about anything that is not clear

You can take a copy of this consent form, to keep. Feel free to take your time thinking about whether you would like to participate. You may wish to discuss your decision with family or friends. Do not sign this consent form unless you have had a chance to ask questions and get answers that make sense to you. By signing this form you will not give up any legal rights.

A description of this clinical trial will be available on http://www.ClinicalTrials.gov, as required by U.S. law. This Web site will not include information that can identify you. At most the Web site will include a summary of the results. You can search this Web site at any time.

#### What is the purpose of this study?

The purpose of this study is to establish the activity of pembrolizumab against cutaneous (skin) squamous cell carcinoma. You have squamous cell cancer from the skin that is no longer curable by surgery or radiation. Previous studies have not established a treatment, such as chemotherapy, that prolongs survival from this disease. Therefore, this study will evaluate whether this drug will shrink the cancer better than previously used treatments such as chemotherapy. Approximately 29 patients will be enrolled on this study.

## What will I be asked to do?

## **Procedures**

If you take part in the study, you will need to do the following:

- Follow the instructions of the study doctor and study staff.
- Take the medicine according to the instructions of the study doctor and the study staff.
- Keep your study appointments. If you must miss one, please contact the study doctor and/or study staff to reschedule as soon as possible.
- Tell the study doctor and/or study staff about any side effects, doctor visits or hospitalizations that you might have had. Tell them about any medication you have been taking, including over the counter and herbal medicines and vitamins and any changes in your usual treatment since your previous visit.
- Inform your study doctor and/or the study staff immediately if you plan to have another medical or surgical treatment. They will discuss with you if this could affect your participation in this study.
- While participating in this study, you should not participate in any other investigational research study.

immediately and discuss with them arrangements for your continuing care.

Approximately 2 tablespoons of blood will also be taken for research purposes.

Study No.: IRB00087412

If you change your mind about participating in this study, please inform the study doctor and/or the study staff

Document Approved On: 9/11/2019

Prior to the start of treatment, you will undergo standard of care procedures to ensure it is safe and feasible to do this study. This will include laboratory studies, imaging such as CT scan or MRI, and a physical examination by your physician. In addition, a biopsy measuring approximately 8 millimeters (0.31 inches) of both normal skin and of your tumor will be performed prior to treatment for research purpose. One to two stitches may be required at time of biopsy.

Once on treatment, you will receive the study drug, pembrolizumab, via a vein once every three weeks. Pembrolizumab will be free of charge. Prior to each treatment you will have laboratory studies drawn and an evaluation including physical exam by your treating physician. These tests are considered standard of care. After 4 treatments (3 months), if feasible, you will undergo repeat biopsy of both normal skin at tumor each measuring approximately 8 mm in size. One to two stitches may be required at time of biopsy. Imaging to evaluate the state of the cancer will be done every 3 months to establish whether the treatment is working. In addition, approximately 2 tablespoons of blood will be drawn for research purposes every three weeks until the 5th dose of treatment.

You will continue on treatment as long as you are not experiencing any undue side effects and as long as your cancer remains stable or shrinks. You can choose to stop the study at any time as well.

As an optional study you may volunteer to have a biopsy of both normal skin and tumor once you discontinue the treatment. The biopsy specimens will be stored for up to 5 years and will be used for future cancer research studies. We will ask if you can follow up with your physician approximately one month after discontinuing treatment to make sure that you have fully recovered from the treatment.

## How will my medicine be provided?

The medicine that you will take will be dispensed by the investigational drug pharmacy and administered to you via a vein in your arm. If you have questions about the medicine, you should ask the principal investigator or study nurse.

## Who owns my study information and samples?

If you join this study, you will be donating your samples and study information. Additional tumor and blood samples will be obtained and used for medical research by the investigators of this study. These samples are valuable to medical research and may help identify a marker to help with the treatment of this disease. The samples are coded to protect your identity. Samples will not be sold or used directly for the production of commercial products.

You are able to request that your tissue/blood samples be destroyed if you change your mind at a later date.

You will not receive any compensation if your samples or information are used to make a new product. If you withdraw from the study, data and samples that were already collected may be still be used for this study. If you ask that your samples not be used, then we will destroy any samples that were previously taken.

### What are the possible risks and discomforts?

Pembrolizumab, which is approved in the USA and some other countries, is available by prescription to treat several different cancers, but may not be approved to treat your type of cancer.

Overall, as of 03-Mar-2018, approximately 25,519 patients have been treated with pembrolizumab in clinical studies.

Pembrolizumab works by helping your immune system to fight your cancer.

However, pembrolizumab can also cause your immune system to attack normal organs and tissues in your body and can affect the way they work, which can result in side effects. These side effects may be serious (i.e. causing hospitalization or be life-threatening), may result in death, and/or may occur after you stop taking pembrolizumab.

#### **Risks and Discomforts**

#### **Pembrolizumab**

PI: Ragini R. Kudchadkar, MD Protocol #: Winship 3185-16

Version Date: 04/15/2019 Page 3 of 13 IRB Form 01292016

Emory University IRB IRB use only

Study No.: IRB00087412

Document Approved On: 9/11/2019

The study doctor believes that the following side effects may be caused by pembrolizumab.

#### **VERY COMMON**

Out of 100 people who receive pembrolizumab, 20 or more people may have the following:

- Itching of the skin
- Loose or watery stools
- Cough

#### COMMON

Out of 100 people who receive pembrolizumab, at least 5 but less than 20 people may have the following:

- Joint Pain
- Rash
- Fever
- · Back pain
- · Pain in your belly
- · Loss of skin color
- Not enough thyroid hormone you may feel tired, gain weight, feel cold, have infrequent or hard stools
- Low level of salt in the blood that may cause you to feel tired, confused, headache, muscle cramps or sick to your stomach

#### **UNCOMMON**

Out of 100 people who receive pembrolizumab, at least 1 but less than 5 people may have the following:

- Inflammation of the lungs so you may feel short of breath and cough. Sometimes this might lead to death
- Too much thyroid hormone so you may feel anxious, angry, have trouble sleeping, feel weak, tremble, sweat, feel tired, have loose and watery stools
- Infusion reaction, where you may feel dizzy or faint, flushed, get a rash, have a fever, feel short of breath at the time of receiving your infusion (IV) or just after, or pain at the site of infusion
- Inflammation of the bowels/gut, which may cause severe pain in your belly with loose or watery stools, and black, tarry, sticky stools or stools with blood or mucus
- Inflammation of the skin so you may have peeling of the skin, itchiness, and/or skin redness. The skin inflammation (i.e. peeling, itching and redness) could also be widespread throughout your body. More severe skin reactions may involve the inside of your mouth, the surface of your eye and genital areas, and/or may cause the top layer of your skin to peel from all over your body which can cause severe infection.

#### **RARE**

## Out of 100 people who receive pembrolizumab, less than 1 person may have the following:

- Inflammation of the nerves that may cause pain, weakness or tingling in your hands and feet, and may spread to your legs, arms and upper body leading to severe muscle weakness and possible temporary paralysis
- Inflammation of the muscles so you may feel weak or have pain in your muscles
- Inflammation of the pancreas (a gland in your abdomen that controls sugar levels) so you may have severe pain in the top part of your belly that may move to your back, feel sick to your stomach, and vomiting that gets worse when you eat
- Inflammation of the eye so you may have eye redness, blurred vision, sensitivity to light, eye pain, see floaters or have headaches
- Inflammation of the liver that may make you feel sick to your stomach and vomit, feel like not eating, feel tired, have a mild fever, have a pain in the right side of your belly, yellow eyes and skin, and dark urine
- Inflammation of the pituitary gland (a gland in the head), which may cause you to feel sick to your stomach or have headaches, changes in your behavior, double vision, few to no menstrual cycles, weakness, vomiting and dizziness or fainting
- Adrenal glands (glands on top of the kidneys) that may not make enough hormone, which could cause tiredness, weight loss, muscle weakness, feeling faint, joint, muscle and belly aches, nausea, vomiting, loose or watery stools, fever, salt craving, and sometimes darkening of the skin like a suntan

• Type 1 Diabetes, a condition that can cause too much sugar in your blood, feeling thirstier than usual, frequent urination and weight loss. You are likely to need regular insulin shots

- Inflammation of the kidney so you may pass less urine or have cloudy or bloody urine, swelling and low back pain
- Inflammation of the middle layer of your heart wall that may cause your heart to have difficulty pumping blood throughout your body, which can cause chest pain, shortness of breath and swelling of the legs. You may experience a fast or irregular heartbeat that may cause dizziness or fainting
- Inflammation of the thyroid gland, an organ that makes and stores thyroid hormones. This condition may lead to change in your heart rate, blood pressure, body temperature, and the rate at which food is converted into energy
- A condition that may make you feel weak and tired and might have drooping of the eyelids, blurred or double vision, difficulty swallowing, slurred speech, weakness in your arms and legs, or difficulty breathing
- The formation of small clusters of immune cells (called granulomas) in parts of your body such as your lymph nodes, eyes, skin, or lungs
- Inflammation of the brain with confusion and fever. This may also include: disorientation, memory problems, seizures (fits), changes in personality and behavior, difficulty speaking, weakness or loss of movement in some parts of your body, and loss of consciousness
- Generalized lipodystrophy which is widespread loss or lack of adipose (fat) tissue leading to muscle weakness, abnormal gait, and impairment in brain function (difficulty speaking, or disorientation).

Additionally, since pembrolizumab was approved in September 2014, the following side effects have been reported by people receiving pembrolizumab. These side effects were voluntarily reported from a group of people of unknown size. It is not possible to estimate the frequency of this side effect:

Inflammation of the joints which may include joint pain, stiffness and/or swelling

**If you have had** an allogeneic stem cell transplant (a procedure in which a person receives blood-forming stem cells from a donor), you may experience graft versus host disease (GvHD), which may include diarrhea, skin rashes, and liver damage, **after receiving pembrolizumab**. Sometimes this condition can lead to death.

If you have had a solid organ transplant (for example, if you have received a kidney or heart transplant), you may experience rejection of the transplanted organ. Your doctor will monitor you and should tell you what signs and symptoms you should report depending on the type of organ transplant that you have had.

Patients treated with pembrolizumab **BEFORE** going on to receive an allogeneic stem cell transplant (a procedure in which a person receives blood-forming stem cells from a donor), should inform their transplant physicians that they have received pembrolizumab in the past.

In patients with any hematologic malignancy (cancers of the blood like Hodgkin lymphoma, multiple myeloma): there is a potential for an increased risk of severe complications following allogeneic stem cell transplant in patients who previously received pembrolizumab **BEFORE** an allogeneic stem cell transplant.

Reports of clotting of blood within the liver and severe graft versus host disease (which can include skin, liver and gastrointestinal symptoms), including death, have been received for patients who received pembrolizumab **BEFORE** an allogeneic stem cell transplant.

## What effects could the tests have on me?

You may feel discomfort during some of these tests or may experience some inconveniences. Some may also have risks, which may include:

Blood samples: drawing blood from your arm may cause pain, bruising, lightheadedness, and rarely, infection.

IV line: may cause discomfort, irritation, mild bruising, bleeding, leakage of drug solution, and rarely, infection, nausea, and lightheadedness. Because pembrolizumab is an antibody, there is the possibility that you may experience an acute

Document Approved On: 9/11/2019

infusion reaction. These are side effects that develop during or immediately after the administration of pembrolizumab signs and symptoms may include:

Document Approved On: 9/11/2019

Version Date: 04/15/2019

IRB Form 01292016

- Blood pressure changes (increase or decrease)
- Cough
- Dizziness
- Fast heart beat
- Feeling cold
- Feeling that the tongue is swelling or your airway is closing and you have trouble breathing
- Fever
- Headache
- Joint pains
- Muscle pains
- Nausea
- Rash, hives, or itching
- Shortness of breath
- Sweating
- Tiredness
- Vomiting

Magnetic resonance imaging, also called MRI scans, use a strong magnetic field. You will be placed in a narrow cylinder, and this could make you feel claustrophobic. The magnetic field can move or alter any solid metal that you have in your body (e.g. pacemaker, artificial valves, joint replacements, cochlear implants or other medical devices). You should mention any such procedures you have had in the past to your doctors to determine whether there might be a risk from an MRI. If you have worked with metal in the past, you also should discuss the specifics with your doctor. An x-ray may be necessary to see whether there is metal left in your body.

Computerized tomography, CT scans are used to create images of internal bones and organs using radiation. High dose radiation is known to produce cancer cells. The effect of exposure to radiation adds up over a lifetime. The amount of radiation exposure involved in this trial will not be significantly greater than for subjects with your disease who do not take part in the trial. The contrast solution that may be given for a CT scan may cause an allergic reaction (rare). Severe allergic reactions can be life threatening. CT contrast solution can cause kidney damage, especially if you are diabetic, dehydrated (lost body water) or elderly.

### Are there any other risks?

Other less common side effects have been reported with the use of the drugs in this study. The study doctor or staff can discuss these with you.

There may be other side effects or risks that are not known at this time.

#### Radiation-Related Risks

You will be exposed to radiation from CT scans. These procedures are necessary for your medical care and will occur even if you do not participate in this study. The radiation dose estimate that you will receive is equal to or less than the radiation exposure allowed to be received by a radiation worker for 5 years. The principal risk associated with a radiation dose is the possibility of developing a radiation-induced cancer later in life. Although the risk from radiation is cumulative it is not expected to adversely affect your condition or treatment. The Emory University Radiation Safety Committee has reviewed and approved the use of radiation in this research study.

## Risks of biopsies

Common side effects of a biopsy are a small amount of bleeding at the time of the procedure, pain at the biopsy site, bruising, swelling and scarring. Rarely, an infection can occur.

## **Pregnancy Risks**

Document Approved On: 9/11/2019

It is not known if the study drug may affect an unborn or nursing baby. If you are pregnant, trying to become pregnant or breast-feeding, you may not be in the study. Non-pregnant, non-breast-feeding women may only be enrolled if they are willing to follow the guidance outlined below, or are considered to be highly unlikely to conceive. Highly unlikely to conceive is defined as 1) surgically sterilized, or 2) postmenopausal (a woman who is 45 years of age or older and has not had menses for greater than

1 year will be considered postmenopausal), or 3) not heterosexually active for the duration of the study.

If you are a woman: to protect against possible side effects of the study drug, women who are pregnant or nursing a child may not take part in this study. If you become pregnant, there may be risks to you, the embryo, or fetus. These risks are not yet known. If you are a woman of childbearing ability, you and the study doctor must agree on a method of birth control to use throughout the study. If you think that you have gotten pregnant during the study, you must tell the study doctor immediately. Pregnant women will be taken out of the study.

**If you are a man:** the effect of the study drug on sperm is not known. To protect against possible side effects, if you are a man you should not get a sexual partner pregnant while taking the study drug and for 180 days after the last dose. You and the study doctor should agree on a method of birth control to use throughout the study.

Patients should use birth control methods that can achieve a failure rate of less than 1% per year when used consistently and correctly and are considered as highly effective birth control methods. Such methods include:

- Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation:
  - Oral
  - Intravaginal
  - Transdermal
- Progestogen-only hormonal contraception associated with inhibition of ovulation:
  - Oral
  - Injectable
  - Implantable
- Intrauterine device (IUD)
- Intrauterine hormone-releasing system (IUS)
- Bilateral tubal occlusion
- Vasectomized partner
- Sexual abstinence

Patients should start using birth control from study Visit 1 throughout the study period up to 180 days after the last dose of study therapy.

If you or your partner become pregnant during the study or within 120 days after stopping the treatment, you should immediately inform your study doctor and/or the study staff (see contact information on first page of this document). If you become pregnant during the study, the study drug will be stopped and you will be taken out of the study.

It is possible that the researchers will learn something new during the study about the risks of being in it. If this happens, they will tell you about it. Then you can decide if you want to continue to be in this study or not. You may be asked to sign a new consent form that includes the new information if you decide to stay in the study.

## Will I benefit directly from the study?

This study is not designed to benefit you directly. Your cancer may improve while you are in this study but it may not, and it may even get worse. This study is designed to learn more about how affective this treatment is for squamous cell cancer from the skin. The study results may be used to help others in the future.

### Will I be compensated for my time and effort?

You will not be offered compensation for being in this study.

What are my other options?

If you decide not to enter this study, there is care available to you outside of the

If you decide not to enter this study, there is care available to you outside of this research study. Option for treatment of your disease is primarily chemotherapy. Please discuss with your physician all the specific chemotherapy drugs that you could potentially be treated with outside of this study.

Taking part in this study, however, may make you unable to participate in some other research studies, if they exclude people who have taken certain treatments. You should discuss this with the researchers if you have concerns. You may wish to research other study options at websites like clinicaltrials.gov and ResearchMatch.org.

## How will you protect my private information that you collect in this study?

Whenever possible, a study number, rather than your name, will be used on study records. Your name and other identifying information will not appear when we present or publish the study results.

Study records can be opened by court order. They also may be provided in response to a subpoena or a request for the production of documents.

## Storing and Sharing your Information

Your samples, genomic data and health information will be stored and shared with other researchers. The samples and information will be available for any research question, such as research to understand what causes certain diseases (for example heart disease, cancer, or psychiatric disorders), development of new scientific methods, or the study of where different groups of people may have come from.

## How is my Genetic Information Protected? What are the Risks?

The Genetic Information Nondiscrimination Act (GINA) is a federal law that generally makes it illegal for health insurance companies, group health plans, and most employers to discriminate against you based on your genetic information. This law generally will protect you in the following ways:

- Health insurance companies and group health plans may not request your genetic information that we get from this research.
- Health insurance companies and group health plans may not use your genetic information when making decisions regarding your eligibility or premiums.
- Employers with 15 or more employees may not use your genetic information that we get from this research when making a decision to hire, promote, or fire you or when setting the terms of your employment.

Be aware that GINA does <u>not</u> protect you against genetic discrimination by companies that sell life insurance, disability insurance, or long-term care insurance, and does not apply to employers with less than 15 employees.

In addition to GINA, the State of Georgia has laws that prohibit insurers from using genetic testing information for any non-treatment purpose. However, like GINA, this state law protection has exclusions: life insurance policies, disability income policies, accidental death or dismemberment policies, Medicare supplement policies, long-term care insurance policies, credit insurance policies, specified disease policies, hospital indemnity policies, blanket accident and sickness policies, franchise policies issued on an insurance policy written as a part of workers' compensation equivalent coverage, or other similar limited accident and sickness policies.

## **Privilege**

In the State of Georgia, your genetic information has special legal protections called "privilege," which means that the information cannot be used as evidence in a court. By signing this form and allowing us to use and disclose your genetic information for the purposes described in this consent, you waive any privilege with regard to that genetic information, meaning that the information loses this legal protection.

## **Medical Record**

If you have been an Emory Healthcare patient before, then you already have an Emory Healthcare medical record. If you have never been an Emory Healthcare patient, you do not have one. An Emory Healthcare medical record will be made for you if an Emory provider or facility gives you any services or procedures for this study.

Emory Healthcare may create study information about you that can help with your care. For example, the results of study tests or procedures. These study results will be put in your Emory Healthcare medical record. Anyone who has access to your medical records will be able to have access to all the study information placed there. The confidentiality of the study

Document Approved On: 9/11/2019

**Emory University IRB** 

Study No.: IRB00087412 IRB use only

information in your medical record will be protected by laws like the HIPAA privacy rule. State and federal laws may not protect the research information from disclosure.

Document Approved On: 9/11/2019

Version Date: 04/15/2019

IRB Form 01292016

The results of some study tests and procedures will be used only for research purposes and will not be placed in your medical record. For this study, those items include:

Research blood work Tumor biopsy Skin biopsy PDL1 testing

Tests and procedures done at non-Emory places may not become part of your Emory medical record. Also, if you decide to be in this study, it is up to you to let your other health providers know.

## In Case of Injury

If you get ill or injured from being in the study, Emory will help you to get medical treatment. Emory and the sponsor have not, however, set aside any money to pay you or to pay for this medical treatment. The only exception is if it is proven that your injury or illness is directly caused by the negligence of an Emory or sponsor employee. "Negligence" is the failure to follow a standard duty of care.

If you become ill or injured from being in this study, your insurer will be billed for your treatment costs. If you do not have insurance, or if your insurer does not pay, then you will have to pay these costs.

If you believe you have become ill or injured from this research, you should contact Dr. Ragini Kudchadkar at telephone . You should also let any health care provider who treats you know that you are in a research study. number

### Costs

The study sponsor will pay for certain items and services that you may receive if you take part in this study. Research specific items will be covered by the study supporter including pembrolizumab, research biopsies and research blood draws.

You will have to pay for the items or services for which the study sponsor does not pay. The sponsor will not pay for your regular medical care. If you have insurance, Emory will submit claims to your insurance for items and services that the sponsor does not cover. Emory will send in only those claims for items and services that it reasonably believes your insurance will pay and that the sponsor has not paid.

The actual amount that you have to pay depends on whether or not you have health insurance and whether or not that insurance will pay for any research study costs. Generally, insurance companies will not pay for items and services that are required just for a research study. Some insurance companies will not pay for regular medical treatment or treatment for complications if you are in a study. How much you will have to pay for any co-payments, deductibles or co-insurance depends on your plan. Emory and the sponsor will not pay for these costs.

It is a good idea to contact your insurance provider and tell them you want to be in this research study. Ask them what they will pay for and what they will not pay for. You can also ask the study team for help in figuring out what you will have to pay.

If you do not have insurance, Emory will review your case as part of its program for low-income patient care. The standard policies of that program will apply. The program will figure out if you have to pay any costs for taking part in the study and what those costs will be.

## Withdrawal from the Study

You have the right to leave a study at any time without penalty.

For your safety, however, you should consider the study doctor's advice about how to go off the study treatment. If you leave the study before the final planned study visit, the researchers may ask you to have some of the final steps done.

Document Approved On: 9/11/2019

The researchers also have the right to stop your participation in this study without your consent for any reason, especially if they believe it is in your best interest or if you were to object to any future changes that may be made in the study plan.

#### Authorization to Use and Disclose Protected Health Information

The privacy of your health information is important to us. We call your health information that identifies you, your "protected health information" or "PHI." To protect your PHI, we will follow federal and state privacy laws, including the Health Insurance Portability and Accountability Act and regulations (HIPAA). We refer to all of these laws as the "Privacy Rules." Here we let you know how we will use and disclose your PHI for the study.

## **Main Study**

## PHI that Will be Used/Disclosed:

The PHI that we will use or share for the main research study includes:

- Medical information about you including your medical history and present/past medications.
- Results of exams, procedures and tests you have before and during the study.
- Laboratory test results.

## Purposes for Which Your PHI Will be Used/Disclosed:

We will use and share your PHI for the conduct and oversight of the research study. We will use and share your PHI to provide you with study related treatment and for payment for such treatment. We will also use and share your PHI to conduct normal business operations. We may share your PHI with other people and places that help us conduct or carry out the study, such as laboratories, data management centers, data monitors, contract research organizations, Institutional Review Boards (IRBs) and other study sites. If you leave the study, we may use your PHI to determine your health, vital status or contact information.

## Use and Disclosure of Your Information That is Required by Law:

We will use and disclose your PHI when we are required to do so by law. This includes laws that require us to report child abuse or abuse of elderly or disabled adults. We will also comply with legal requests or orders that require us to disclose your PHI. These include subpoenas or court orders.

#### Authorization to Use PHI is Required to Participate:

By signing this form, you give us permission to use and share your PHI as described in this document. You do not have to sign this form to authorize the use and disclosure of your PHI. If you do not sign this form, then you may not participate in the research study or receive research-related treatment. You may still receive non-research related treatment.

## People Who will Use/Disclose Your PHI:

The following people and groups will use and disclose your PHI in connection with the research study:

- The Principal Investigator and the research staff will use and disclose your PHI to conduct the study and give you study related treatment.
- Emory may use and disclose your PHI to get payment for study related treatment and to run normal business operations.
- The Principal Investigator and research staff will share your PHI with other people and groups to help conduct the study or to provide oversight for the study.
- Ragini R. Kudchadkar, MD is the Sponsor of the study. The Sponsor may use and disclose your PHI to
  make sure the research is done correctly and to collect and analyze the results of the research. The
  Sponsor may disclose your PHI to other people and groups like study monitors to help conduct the study
  or to provide oversight for the study.
- The following people and groups will use your PHI to make sure the research is done correctly and safely:

Version Date: 04/15/2019

IRB Form 01292016

Study No.: IRB00087412 Emory Ur

## Emory University IRB IRB use only

 Emory offices that are part of the Human Research Participant Protection Program and those that are involved in study administration and billing. These include the Emory IRB, the Emory Research and Healthcare Compliance Offices, and the Emory Office for Clinical Research.

Document Approved On: 9/11/2019

Version Date: 04/15/2019

IRB Form 01292016

- o Government agencies that regulate the research including: Food and Drug Administration
- Public health agencies
- o Research monitors and reviewer.
- o Accreditation agencies.
- Merck- study drug manufacturer
- Sometimes a Principal Investigator or other researcher moves to a different institution. If this happens,
  your PHI may be shared with that new institution and their oversight offices. PHI will be shared securely
  and under a legal agreement to ensure it continues to be used under the terms of this consent and HIPAA
  authorization.

Optional Study Skin and cancer biopsy after discontinuing the treatment:

PHI That Will be Used/Disclosed for Optional Study:

The PHI that we will use and/or disclose (share) for the optional research study includes:

- Medical information about you including your medical history and present/past medications.
- Results of exams, procedures and tests you have before and during the study.
- Laboratory test results.

Purposes for which your PHI will be Used/Disclosed for Optional Study:

We will use and disclose your PHI for the conduct and oversight of the optional research study, including the administration and payment of any costs relating to subject injury.

Authorization for This Use of PHI is Required to Participate in Optional Study, but Not in Main Study: You do not have to authorize the use and disclosure of your PHI. If you do not authorize the use and disclosure of your PHI for the optional study, then you may not participate in the optional research study. You can still be in the main research study even if you don't participate in the optional study.

People Who Will Use/Disclose Your PHI for Optional Study:

The following people and groups will use and disclose your PHI in connection with the optional research study:

• The same people and groups who will use and disclose your PHI for the Main Study will also do so in connection with the optional research study/storage of PHI for future research

## **Revoking Your Authorization**

If you sign this form, at any time later you may revoke (take back) your permission to use your information. If you want to do this, you must contact the study team at: Dr. Ragini Kudchadkar at

At that point, the researchers would not collect any more of your PHI. But they may use or disclose the information you already gave them so they can follow the law, protect your safety, or make sure that the study was done properly and the data is correct. If you revoke your authorization you will not be able to stay in the study.

### Other Items You Should Know about Your Privacy

Not all people and entities are covered by the Privacy Rules. HIPAA only applies to health care providers, health care payers, and health care clearinghouses. If we disclose your information to people who are not covered by the Privacy Rules, including HIPAA, then your information won't be protected by the Privacy Rules. People who do not have to follow the Privacy rules can use or disclose your information with others without your permission if they are allowed to do so by the laws that cover them.

To maintain the integrity of this research study, you generally will not have access to your PHI related to this research until the study is complete. When the study ends, and at your request, you generally will have access to your PHI that we maintain in a designated record set. A designated record set is data that includes medical information or billing records that your health care providers use to make decisions about you. If it is necessary for your health care, your health information will be provided to your doctor.

# **Emory University IRB**

Study No.: IRB00087412 Document Approved On: 9/11/2019 IRB use only

We may remove identifying information from your PHI. Once we do this, the remaining information will not be subject to the Privacy Rules. Information without identifiers may be used or disclosed with other people or organizations for purposes besides this study.

## **Contact Information**

Contact Dr. Ragini Kudchadkar at

- if you have any questions about this study or your part in it,
- if you feel you have had a research-related injury or a bad reaction to the study drug, or
- if you have questions, concerns or complaints about the research

Contact the Emory Institutional Review Board at

- if you have guestions about your rights as a research participant.
- if you have questions, concerns or complaints about the research.
- You may also let the IRB know about your experience as a research participant through our Research Participant Survey at http://www.surveymonkey.com/s/6ZDMW75.

Version Date: 04/15/2019 IRB Form 01292016

**Emory University IRB** 

## IRB use only

## **Consent and Authorization** Consent and HIPAA Authorization for Optional Study/Studies: Please initial below if you opt to participate in and authorize use and disclosure of your PHI in the optional study/studies previously described: Skin and cancer biopsy after discontinuing the treatment Initials TO BE FILLED OUT BY SUBJECT ONLY Please print your name, sign, and date below if you agree to be in the main study. By signing this consent and authorization form, you will not give up any of your legal rights. We will give you a copy of the signed form to keep.

Document Approved On: 9/11/2019

Version Date: 04/15/2019

IRB Form 01292016

#### am / pm Signature of Subject (18 years or older and able to consent) Date Time (please circle)

TO BE FILLED OUT BY STUDY TEAM ONLY

## Name of Person Conducting Informed Consent Discussion am / pm **Signature of Person Conducting Informed Consent Date** Time (please circle) Discussion

Study No.: IRB00087412

Name of Subject